CLINICAL TRIAL: NCT02531594
Title: An Intervention to Reduce Second Hand Smoke Exposure Among Pediatric Emergency Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CINC 2015-1914; 1R01HD083354 (NIH); R01ES027815 (NIH)
Record Dates: First submitted 2015-08-04; First posted 2015-08-24 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBIRT (Experimental): An assessment form, motivational interviewing, personalized educational materials, immediate access to cessation resources, a 12-week supply of nicotine replacement therapy and weekly booster materials for 12 weeks.
  nicotine
  Interventions: Behavioral: SBIRT
- HHC (Placebo Comparator): The Healthy Habits Control program has been previously developed and used in the out-patient setting, and will be used as an attention control in which caregivers will receive instruction on healthy lifestyle choices to improve their child's health. Cessation assistance will be offered at the study's conclusion.
  Interventions: Behavioral: HHC

INTERVENTIONS:
Behavioral: SBIRT — The Social Worker will provide caregivers with the brief (10-15 minute) "Advise, Assess, Assist" intervention based on the Clinical Practice Guidelines, and tailored on levels of motivation to quit and tobacco dependence. Patients in this group will receive Nicotine Replacement Therapy vouchers, immediate connection to cessation resources, and intervention materials.
  Arms: SBIRT
Behavioral: HHC — The Social Worker will provide caregivers with the brief (10-15 minute) "Lets Go! 5-2-1-0" intervention which is a child obesity prevention program. Patients in this group will receive motivational interviewing in regards to helping children and families eat healthy and be active. This group will receive water bottle vouchers, immediate connection to 5-2-1-0 resources, and intervention materials.
  Arms: HHC

SUMMARY:
This study will test the efficacy of a cessation intervention for caregivers in a large, inner-city Pediatric Emergency Department. The investigators will randomize 750 caregivers who smoke who present to our Pediatric Emergency Department with their child who has a Second Hand Smoke exposure-related illness to either one of two conditions: 1) Screening, Brief Intervention, and Assisted Referral to Treatment (SBIRT); or 2) Healthy Habits Control (HHC). The Screening, Brief Intervention, and Assisted Referral to Treatment condition will include a brief form of the Clinical Practice Guideline: Treating Tobacco Use and Dependence, motivational interviewing, engaging and personalized materials on the effects of smoking and Second Hand Smoke exposure, immediate access to caregivers' choice of cessation resources (e.g., Quitline, smokefree.gov, or txt2quit), a 12-week supply of nicotine replacement therapy and weekly booster materials for 12 weeks. The Healthy Habits Control program will be used as an attention control in which caregivers will receive instruction on healthy lifestyle choices to improve the child's health.

DETAILED DESCRIPTION:
This study will test the efficacy of a cessation intervention for caregivers in a large, inner-city Pediatric Emergency Department. The proposed Screening, Brief Intervention, and Assisted Referral to Treatment will highlight the effects of Second Hand Smoke exposure on the child's health. the investigators will randomize 750 caregivers who smoke who present to our Pediatric Emergency Department with their child who has a Second Hand Smoke exposure related illness to either one of two conditions: 1) Screening, Brief Intervention, and Assisted Referral to Treatment; or 2) Healthy Habits Control. The Screening, Brief Intervention, and Assisted Referral to Treatment condition will use components shown to be effective in the out-patient setting but not yet tested in the Pediatric Emergency Department setting. It will include a brief form of the Clinical Practice Guideline: Treating Tobacco Use and Dependence, motivational interviewing, engaging and personalized materials on the effects of smoking and Second Hand Smoke exposure, immediate access to caregivers' choice of cessation resources (e.g., Quitline, smokefree.gov, or txt2quit), a 12-week supply of nicotine replacement therapy and weekly booster materials for 12 weeks. The Healthy Habits Control program has been previously developed and used in the out-patient setting, and will be used as an attention control in which caregivers will receive instruction on healthy lifestyle choices to improve their child's health. Cessation assistance will be offered at the study's conclusion. If effective, the Screening, Brief Intervention, and Assisted Referral to Treatment model could be routinely used in the Pediatric Emergency Department setting, which could reach at least one million smokers a year, and could result in significant reductions in caregivers' tobacco use, Second Hand Smoke exposure related pediatric illness, and costs in this population. In addition, the investigators' results will inform the conduct of public health research efforts aimed at adults via the Pediatric Emergency Department.

ELIGIBILITY:
Inclusion Criteria:Eligible participants must:

1. be > age 18;
2. be accompanying a child 0-17 years of age who is presenting to the Pediatric Emergency Department with:

   * a stable condition, that is, patients who are not critically ill and do not require immediate treatment and intervention by the Pediatric Emergency Department practitioner and
   * a potentially Second Hand Smoke exposure related chief complaint (such as wheezing, difficulty breathing, cough) as outlined by the U.S. Surgeon General;45
3. be a daily smoker;
4. have currently or recently smoked inside their home;
5. speak and read English, and
6. have a permanent address and a working cell or landline number.
7. Live within a 50 mile radius.
8. Child is a non-smoker.

Exclusion Criteria: Caregivers will be excluded if

1. their child has a tracheostomy or
2. if the caregivers are tobacco chewers only,
3. if the caregivers are using pharmacologic cessation treatment,
4. or plan to move within the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Melinda Mahabee-Gittens, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahabee-Gittens EM, Ammerman RT, Khoury JC, Stone L, Meyers GT, Witry JK, Merianos AL, Mancuso TF, Stackpole KMW, Bennett BL, Akers L, Gordon JS. Healthy families: study protocol for a randomized controlled trial of a screening, brief intervention, and referral to treatment intervention for caregivers to reduce secondhand smoke exposure among pediatric emergency patients. BMC Public Health. 2017 May 2;17(1):374. doi: 10.1186/s12889-017-4278-8. PMID 28464887
- [Result] Mahabee-Gittens EM, Ammerman RT, Khoury JC, Tabangin ME, Ding L, Merianos AL, Stone L, Gordon JS. A Parental Smoking Cessation Intervention in the Pediatric Emergency Setting: A Randomized Trial. Int J Environ Res Public Health. 2020 Nov 4;17(21):8151. doi: 10.3390/ijerph17218151. PMID 33158230
- [Result] Mahabee-Gittens EM, Merianos AL, Fulkerson PC, Stone L, Matt GE. The Association of Environmental Tobacco Smoke Exposure and Inflammatory Markers in Hospitalized Children. Int J Environ Res Public Health. 2019 Nov 21;16(23):4625. doi: 10.3390/ijerph16234625. PMID 31766400
- [Result] Mahabee-Gittens EM, Merianos AL, Stone L, Tabangin ME, Khoury JC, Gordon JS. Tobacco Use Behaviors and Perceptions of Parental Smokers in the Emergency Department Setting. Tob Use Insights. 2019 Jun 19;12:1179173X19841392. doi: 10.1177/1179173X19841392. eCollection 2019. PMID 31258335
- [Result] Mahabee-Gittens EM, Merianos AL, Tabangin ME, Stone L, Gordon JS, Khoury JC. Provision of free nicotine replacement therapy to parental smokers in the pediatric emergency setting. Tob Prev Cessat. 2020 May 18;6:30. doi: 10.18332/tpc/119125. eCollection 2020. PMID 32760865
- [Result] Mahabee-Gittens EM, Mazzella MJ, Doucette JT, Merianos AL, Stone L, Wullenweber CA, A Busgang S, Matt GE. Comparison of Liquid Chromatography Mass Spectrometry and Enzyme-Linked Immunosorbent Assay Methods to Measure Salivary Cotinine Levels in Ill Children. Int J Environ Res Public Health. 2020 Feb 12;17(4):1157. doi: 10.3390/ijerph17041157. PMID 32059566
- [Derived] Mahabee-Gittens EM, Matt GE, Hoh E, Quintana PJE, Stone L, Geraci MA, Wullenweber CA, Koutsounadis GN, Ruwe AG, Meyers GT, Zakrajsek MA, Witry JK, Merianos AL. Contribution of thirdhand smoke to overall tobacco smoke exposure in pediatric patients: study protocol. BMC Public Health. 2019 May 2;19(1):491. doi: 10.1186/s12889-019-6829-7. PMID 31046729
- [Derived] Mahabee-Gittens EM, Merianos AL, Matt GE. Preliminary evidence that high levels of nicotine on children's hands may contribute to overall tobacco smoke exposure. Tob Control. 2018 Mar;27(2):217-219. doi: 10.1136/tobaccocontrol-2016-053602. Epub 2017 Mar 30. PMID 28360145

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The numbers listed below represent a dyad (child participant/caregiver participant).
Groups:
- SBIRT: An assessment form, motivational interviewing, personalized educational materials, immediate access to cessation resources, a 12-week supply of nicotine replacement therapy and weekly booster materials for 12 weeks.
  nicotine
  SBIRT: The Social Worker will provide caregivers with the brief (10-15 minute) "Advise, Assess, Assist" intervention based on the Clinical Practice Guidelines, and tailored on levels of motivation to quit and tobacco dependence. Patients in this group will receive Nicotine Replacement Therapy vouchers, immediate connection to cessation resources, and intervention materials.
- Healthy Habits Control: The Healthy Habits Control program has been previously developed and used in the out-patient setting, and will be used as an attention control in which caregivers will receive instruction on healthy lifestyle choices to improve their child's health. Cessation assistance will be offered at the study's conclusion.
  HHC: The Social Worker will provide caregivers with the brief (10-15 minute) "Lets Go! 5-2-1-0" intervention which is a child obesity prevention program. Patients in this group will receive motivational interviewing in regards to helping children and families eat healthy and be active. This group will receive water bottle vouchers, immediate connection to 5-2-1-0 resources, and intervention materials.
Period: Overall Study
Arm/Group | SBIRT | Healthy Habits Control
Started | 384 (This represents a dyad (child participant/caregiver participant).) | 381 (This represents a dyad (child participant/caregiver participant).)
Completed | 377 (This represents a dyad (child participant/caregiver participant).) | 373 (This represents a dyad (child participant/caregiver participant).)
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 7 | 8

BASELINE CHARACTERISTICS:
Population: These numbers represent child/caregiver dyads. There were 5 participants who signed consent but withdrew prior to being randomized, thus, the number of participants who signed consent was 770 but the number of participants randomized was 765. Of those, 8 HHC and 7 SBIRT dyads withdrew prior to completing baseline procedures, and therefore were not included in the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Habits Control | SBIRT | Total
Number analyzed (Participants) | 373 | 377 | 750
Age, Categorical [Count of Participants; unit: Participants] — Ages below are reported for the child participants and separately for the caregiver participants. The protocol number enrolled of 770 indicates the number of dyads (child participants/caregiver participants).
  Participants
    Child Participants: <=18 years | 373 | 377 | 750
    Child Participants: Between 18 and 65 years | 0 | 0 | 0
    Child Participants: >=65 years | 0 | 0 | 0
    Caregiver participants: <=18 years | 0 | 0 | 0
    Caregiver participants: Between 18 and 65 years | 373 | 377 | 750
    Caregiver participants: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Measure Description: Ages below are reported for the child participants and separately for the caregiver participants. The protocol number enrolled of 770 indicates the number of dyads (child participants/caregiver participants).
  years
    Child Participants | 4.73 (4.51) | 5.12 (4.89) | 4.92 (4.70)
    Caregiver Participants | 32.59 (7.06) | 33.12 (8.20) | 32.89 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some participants' gender was not reported in baseline questionnaire.
  Participants
    Child Participants: Female | 177 | 185 | 362
    Child Participants: Male | 196 | 192 | 388
    Caregiver Participants: Female | 321 | 330 | 651
    Caregiver Participants: Male | 52 | 47 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Child Participants: Hispanic or Latino | 4 | 8 | 12
  Child Participants: Not Hispanic or Latino | 369 | 368 | 737
  Child Participants: Unknown or Not Reported | 0 | 1 | 1
  Caregiver Participants: Hispanic or Latino | 9 | 8 | 17
  Caregiver Participants: Not Hispanic or Latino | 363 | 368 | 731
  Caregiver Participants: Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Child Participants: American Indian or Alaska Native | 1 | 0 | 1
  Child Participants: Asian | 0 | 1 | 1
  Child Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Child Participants: Black or African American | 215 | 215 | 430
  Child Participants: White | 142 | 137 | 279
  Child Participants: More than one race | 8 | 15 | 23
  Child Participants: Unknown or Not Reported | 7 | 9 | 16
  Caregiver Participants: American Indian or Alaska Native | 2 | 1 | 3
  Caregiver Participants: Asian | 0 | 0 | 0
  Caregiver Participants: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Caregiver Participants: Black or African American | 200 | 200 | 400
  Caregiver Participants: White | 150 | 152 | 302
  Caregiver Participants: More than one race | 18 | 23 | 41
  Caregiver Participants: Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 373 | 377 | 750

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Self-reported Prolonged Abstinence at 6 Weeks
Description: Primary outcomes are self-reported prolonged abstinence at 6-weeks post-enrollment, validated in all participants via salivary cotinine levels.
Time Frame: 6 weeks post enrollment
Measure: Number; unit: percentage of participants
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
percentage of participants | 4.2 | 4.2

2. Primary Outcome: Percentage of Participants With Self-reported Prolonged Abstinence at 6 Months
Description: Primary outcomes are self-reported prolonged abstinence at 6 months post-enrollment, validated in all participants via salivary cotinine levels.
Time Frame: 6months post enrollment
Measure: Number; unit: percentage of participants
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
percentage of participants | 12.9 | 8.3

3. Secondary Outcome: Change From Baseline in the Number of Cigarettes Smoked Per Day at 6 Weeks
Description: Secondary outcomes include number of cigarettes smoked at 6 weeks post enrollment. This number is reporting a change in the number of cigarettes smoked between baseline and six weeks.
Time Frame: baseline and 6 weeks post enrollment
Measure: Median (Inter-Quartile Range); unit: cigarettes per week
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
cigarettes per week | -2 [-5 to 0] | 0 [-4 to 0]

4. Secondary Outcome: Change From Baseline in the Number of Cigarettes Smoked Per Day at 6 Months
Description: Secondary outcomes include number of cigarettes smoked at 6 months post enrollment as compared with baseline.
Time Frame: baseline and 6 months post enrollment
Measure: Median (Inter-Quartile Range); unit: cigarettes per week
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
cigarettes per week | -4 [-9 to -1] | -2 [-5 to 0]

5. Secondary Outcome: Number of Quit Attempts at 6 Weeks
Description: Secondary outcomes include number of quit attempts at 6 weeks post enrollment.
Time Frame: 6 weeks post enrollment
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
quit attempts | 2.69 (5.0) | 2.22 (2.5)

6. Secondary Outcome: Number of Quit Attempts at 6 Months
Description: Secondary outcomes include number of quit attempts at 6 months post enrollment.
Time Frame: 6 months post enrollment
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
quit attempts | 3.82 (6.4) | 2.3 (3.2)

7. Secondary Outcome: Readiness to Quit at 6 Weeks
Description: Secondary outcomes include readiness to quit at 6 weeks post enrollment as measured by a readiness to quit scale.
  Scale name: The Contemplation Ladder Reference: Biener L., Abrams D.B. The Contemplation Ladder: Validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10:360-365. doi: 10.1037/0278-6133.10.5.360.
  What scale measures: the smoker's motivation to quit smoking. The Contemplation Ladder is a validated score that correlates with the likelihood of making a quit attempt and participation in activities associated with quit attempts.
  The Contemplation Ladder is a 1-item, 11-point scale of motivation to quit. The question asks: "Mark the number that shows how you feel about quitting.
  Minimum score: 0 = no thought of quitting Maximum score: 10= taking action to quit Lower scores indicate worse outcomes. Higher scores indicate better outcomes. There are no subscales and one score is chosen by the smoker.
Time Frame: 6 weeks post enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
units on a scale | 6.98 (2.5) | 6.46 (2.8)

8. Secondary Outcome: Readiness to Quit at 6 Months
Description: Secondary outcomes include readiness to quit at 6 months post enrollment as measured by a readiness to quit scale.
  Scale name: The Contemplation Ladder Reference: Biener L., Abrams D.B. The Contemplation Ladder: Validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10:360-365. doi: 10.1037/0278-6133.10.5.360.
  What scale measures: the smoker's motivation to quit smoking. The Contemplation Ladder is a validated score that correlates with the likelihood of making a quit attempt and participation in activities associated with quit attempts.
  The Contemplation Ladder is a 1-item, 11-point scale of motivation to quit. The question asks: "Mark the number that shows how you feel about quitting.
  Minimum score: 0 = no thought of quitting Maximum score: 10= taking action to quit Lower scores indicate worse outcomes. Higher scores indicate better outcomes. There are no subscales and one score is chosen by the smoker.
Time Frame: 6 months post enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
units on a scale | 7.03 (2.6) | 6.77 (2.8)

9. Secondary Outcome: Use of Cessation Resources at 6 Weeks
Description: Secondary outcomes include use of cessation resources at 6 weeks post enrollment.
Time Frame: 6 weeks post enrollment
Measure: Number; unit: Percentage of caregivers
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 377 | 373
Percentage of caregivers | 53 | 0

10. Secondary Outcome: Use of Cessation Resources at 6 Months
Description: Secondary outcomes include use of cessation resources at 6 months post enrollment.
Time Frame: 6 months post enrollment
Population: Data were not collected.
Arm/Group | SBIRT | Healthy Habits Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Six months.
Arm/Group | SBIRT | Healthy Habits Control
All-Cause Mortality (participants affected / at risk) | 0/377 | 0/373
Serious Adverse Events (participants affected / at risk) | 0/377 | 0/373
Other Adverse Events (participants affected / at risk) | 0/377 | 0/373

LIMITATIONS AND CAVEATS:
It should be noted that outcome measure "Use of Cessation Resources at 6 Months" was not reported due to no data being obtained due to lack of resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT02531594/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02531594/ICF_001.pdf